CLINICAL TRIAL: NCT00970411
Title: An Open-label, Non-randomised Dose Escalation Study of KRN951 Administered Orally to Patients With Solid Tumors
Brief Title: Study of KRN951 in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KRN951-001
Record Dates: First submitted 2009-08-31; First posted 2009-09-02 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Solid Tumors
MeSH Terms: interventions — tivozanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- KRN951 (Experimental)
  Interventions: Drug: KRN951

INTERVENTIONS:
Drug: KRN951 — Orally once daily administration

SUMMARY:
The purpose of this study is to assess the safety and tolerability of KRN951 administered to patients with solid tumors. In the single dose period, patients in each cohort will receive one oral dose of KRN951 in the first day, followed by a 6-day rest period during which no treatment is received. After that, patients in each cohort will receive one oral dose of KRN951 daily over a 21-day treatment period, followed by a 7-day rest period during which no treatment is received. Treatment will be continued in the absence of disease progression or unacceptable adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Solid tumors to be unresponsive to, or untreatable by standard therapies
* ≥ three-month life expectancy
* Eastern Cooperative Oncology Group Performance Status score of 0, 1 or 2

Exclusion Criteria:

* Hematologic abnormality
* Myocardial infarction or clinically symptomatic left ventricular failure
* Active hypertension or controllable hypertension more than 3 antihypertensive medications
* Symptomatic CNS metastasis
* Unhealed wounds
* Active infections
* Hepatic or renal functional disorder
* Any of the HBs antigen, HCV antibody and HIV antibody positivity
* Prior use of any chemotherapy, radiotherapy, immunotherapy or surgery within four weeks previous to first dose of study drug
* Pregnant or lactating women
* Women of childbearing potential and fertile men, unless willing to use adequate contraceptive protection

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2009-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
To define the maximum tolerated dose (MTD) of KRN-951 when administered orally for 21 days followed by a 7-day rest period.
To evaluate the safety profile and the tolerability of KRN951 throughout the study period by assessing adverse events and laboratory values recorded during treatment.

SECONDARY OUTCOMES:
To determine the pharmacokinetics of KRN951 in serum
To describe biological and clinical anti-tumor activity

CONTACTS AND LOCATIONS:
Locations (1):
- Shizuoka, Japan